CLINICAL TRIAL: NCT02272296
Title: Reproducibility of Insulin Action When Administered by Needle-free Jet Injection
Brief Title: Reliability of Insulin by Jet Injection
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PKPD_INSJ_4
Record Dates: First submitted 2014-10-14; First posted 2014-10-22 (Estimated); Last update posted 2015-10-28 (Estimated); Status verified 2015-10

CONDITIONS: Diabetes Mellitus
Keywords: Injections, Jet; pharmacology; Insulin Aspart; Equipment and Supplies
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Jet Injector_main study (Active Comparator): Administration of insulin or placebo injection in main study
  Interventions: Device: jet injector; Device: Conventional pen (NovoPen IV)
- conventional pen, NovoPen IV (Placebo Comparator): Administration of insulin or placebo injection in main study
  Interventions: Device: jet injector; Device: Conventional pen (NovoPen IV)
- jet injector_sub study (Active Comparator): Administration of insulin or placebo injection in sub study
  Interventions: Device: jet injector

INTERVENTIONS:
Device: jet injector — 1 administration of insulin in a dose of 0.2 units per kg body weight subcutaneously in the abdomen, 1 empty administration
  Other Names: Insujet™, European Pharma Group, The Netherlands
Device: Conventional pen (NovoPen IV) — 1 administration of insulin in a dose of 0.2 units per kg body weight subcutaneously in the abdomen, 1 empty administration
  Other Names: NovoPen IV, Novo Nordisk
  Arms: Jet Injector_main study; conventional pen, NovoPen IV

SUMMARY:
Using a specific jet injector for the administration of a rapid-acting insulin analogue has been shown to advance the absorption of insulin from the subcutaneous area into the bloodstream by 40-50%, when compared to conventional injection by insulin pens. The reproducibility of the jet stream method has not been previously determined in vivo. It is also unknown how the efficacy of injecting regular insulin by jet stream compares to that of rapid-acting analogues injected by conventional pen.

Objectives: 1. To compare the pharmacologic reproducibility of the rapid-acting insulin analogue aspart (Novorapid®) injected by jet-injection to that of the same insulin injected with a conventional pen. 2. To compare pharmacokinetic and -dynamic profile of regular insulin injected by jet injection to that of aspart insulin injected by conventional pen.

Study design: Double-blind double-dummy randomized controlled parallel/cross-over

DETAILED DESCRIPTION:
1. Introduction Insulin administration by a jet injector is a needle-free alternative to conventional administration of insulin by insulin pens or syringes. Jet injectors deliver insulin at a high velocity (typically >100m/s) across the skin in the subcutaneous tissue and dispense the insulin over a larger area than insulin injected with a syringe. This significantly accelerates absorption of rapid-acting insulin from the subcutaneous area into the systemic circulation.

   Reproducibility of the insulin effect is an essential, but easily overlooked, issue for a product that needs to be administered so frequently in daily practice. When identical doses of aspart insulin were injected by a common syringe on two different days separated by at least a week, the intra-individual and inter-individual variability of various pharmacokinetic and -dynamic parameters was found to vary between 11-21% and 18-36%, respectively. Reproducibility has not been investigated when insulin was administered by jet injectors. The investigators previous studies indicated smaller between-subjects variability in insulin absorption after injection by this jet injector than after injection by conventional pen, providing some evidence that reproducibility is at least comparable, but potentially even better when using a jet injector.

   The aim of the present research proposal is to compare the variability of the metabolic effect of insulin aspart when administered by jet injection to that when injected by conventional insulin pen, under controlled experimental conditions.

   An additional aim is to investigate the pharmacokinetic and -dynamic comparability between regular soluble insulin injected by the jet stream device with aspart insulin administered by conventional pen. The reason the investigators wanted to investigate the comparability is that rapid-acting insulin analogs are not worldwide available and very costly compared to regular insulin. If you could achieve the same pharmacological benefits as rapid acting insulin with a less costly type of insulin, this would be of great benefit for patients with diabetes in less developed countries.
2. Hypotheses The variability of the metabolic effect of insulin administered subcutaneously by jet injection is similar to or better than that of insulin administered by a conventional insulin pen. The investigators also hypothesize that the metabolic effect of soluble insulin administered by jet injection is similar to that of insulin aspart administered by conventional insulin pen.
3. Study Population For this study, a total of 30 healthy volunteers will be recruited. Subjects are potentially eligible when they are between 18 and 50 years of age and in good clinical condition. Additional participants will be recruited in case of drop-out.
4. Investigational medicinal products Main study: Insulin aspart (Novorapid® Penfill 100 units/ml, 3 ml ampoule): rapid-acting analogue of human insulin.

   Sub-study: Regular Human Insulin (Humulin® Penfill 100 units/ml, 3ml ampoule): human regular insulin.
5. Summary of known and potential risks and benefits Novorapid® insulin is indicated for the treatment of diabetes mellitus in adults, adolescents and children above the age of 2 years. The study comprises a risk of hypoglycemia. However, the risk of hypoglycaemia during the experiment is negligible, since glucose is measured at 5-10 minute intervals and additional glucose will be administered should glucose levels tend to drop below 4.8 mmol/l. Intravenous glucose 20% may cause local irritation and occasionally phlebitis.
6. Methods 6.1 Randomisation The study will have a randomised controlled parallel design. Randomisation will be done by a computer program with the use of blocks of two subjects, to randomize which of the two devices will contain insulin and which placebo solution. This will ensure that equal number of subjects will have the experiment with the investigational product (InsujetTM pen) or with the control device (Novopen® IV insulin pen).

   To ensure blinding, both pen devices will be prepared by a nurse who is not otherwise involved in conducting the experiments. There is no indication for prematurely breaking the randomisation code, as subjects will receive the same amount of insulin with one of the two devices in each experiment, with frequent glucose-monitoring to prevent hypoglycemia.

   6.2 Study procedures Potentially eligible study participants will be recruited using websites or by using the RUMC social media. Should this be insufficient, advertisements in local newspapers will be placed. Eligibility will be determined at the screening visit after a medical interview and physical examination.

   Experimental procedures All participants will be examined on two occasions, within 1 week, with one of the two devices containing insulin and the other device as a placebo device.

   Patients will be instructed to consume a low-glycemic index meal the evening before experiments and remain in fasting condition from 20:00 hours onwards.

   On the first and second experimental day, participants will be admitted to the research unit at 08.00 hours in fasting condition and having abstained from smoking, alcohol use and caffeine use for at least 24 hours. A catheter will be inserted in retrograde fashion in a dorsal hand vein for frequent blood sampling, whereby the hand will be placed inside a heated box (air temperature, ~55°C) to arterialize venous blood. Another catheter will be inserted in the antecubital vein of the other arm, which will be kept patent by saline drip, and which will be used for administration of 20% glucose.

   After cannulations, blood will be taken for direct measurement of plasma glucose and stored for later measurement of plasma insulin levels. Thereafter, an independent research nurse will administer insulin at a dose of 0.2 units per kg body weight subcutaneously at the abdominal site, with either the jet injector (InsujetTM) or the conventional pen (Novopen® IV). The device not used for insulin administration will be prepared by the research nurse as well. However, this device is empty although to the patient it will look and feel the same way as the pens filled with insulin. The insulin injection and the simulated injection will be given simultaneously. After injection, the administration site will be covered by the research nurse with a bandage to prevent that the investigator and patient will be able to see whether there has remained some insulin on the skin or not. The investigators as well as the participants will be blinded to which pen contains the insulin and which pen was the placebo device. Subsequently, a 6-hour normoglycemic glucose clamp will be employed, as described previously. To this end, glucose 20% will be administered intravenously at a sufficient rate to maintain normoglycemia, based on plasma glucose levels measured at 5-minute intervals during the first 3 hours and at 10-minute intervals during the remainder of the experiment. Also, blood will be drawn and stored at -80°C every 5 minutes during the first hour after insulin injection and every 15 minutes during the hour thereafter for later determination of plasma insulin and C-peptide levels. During the last four hours, insulin will be measured with 30 minutes intervals. Six hours after the insulin injection, the experiment will be terminated and the patients will be given a meal. The total duration of the study day, including preparation and recovery time, will be 7 hours.

   Participants will be asked separately to return to the research unit a third time for a similar 6-hour normoglycemic glucose clamp. On this occasion, the insulin aspart will be replaced by regular soluble insulin. The insulin will be administered by the jet injector. Pharmacokinetic and -dynamic data obtained from this experiment will be compared with data obtained after injection of aspart insulin by conventional pen both in this study and in a previous investigation.

   The investigators will also ask the subject on both experimental days, within 30 minutes after insulin injection, to point out on a numeric rating scale from 0 to 10 the amount of discomfort or pain and the ease of use experienced with the two administration methods. After the second experiment day, patients will be asked which of the two devices they would prefer for insulin injection, should they have a choice.

   Withdrawal of study subjects Subjects can leave the study at any time for any reason if they wish to do so without any consequences. The investigator can decide to withdraw a subject from the study in case of a severe adverse event or another condition requiring immediate medical care. Appropriate follow up and treatment of withdrawn subjects will be assured. Every subject that withdraws from the study will be replaced with an additional study participant.

   Premature termination of the study The study will be terminated prematurely when unexpected serious adverse events are experienced which endanger other subjects. If the trial is prematurely terminated the investigator will promptly inform the trial subjects, the METC and competent authority. A detailed written explanation of the termination will be provided. Appropriate follow up and treatment of trial subjects will be assured.
7. Safety reporting The investigator will inform the subjects and the reviewing accredited METC if anything occurs, on the basis of which it appears that the disadvantages of participation may be significantly greater than was foreseen in the research proposal. The study will be suspended pending further review by the accredited METC, except insofar as suspension would jeopardise the subjects' health. The investigator will take care that all subjects are kept informed. All (serious) adverse events reported spontaneously by the subject or observed by the investigator or his staff will be recorded and reported at the METC.
8. Statistical analysis Descriptive parameters will be presented as mean ± standard error of the mean. Unpaired T-tests will be performed to compare all main and secondary study endpoints as well as most ease of use and safety endpoints. A Chi2 test will be used to compare the number of patients experiencing post injection hypoglycaemia with the two injection devices. A P-value of < 0.05 will be considered as statistically significant. All statistical analyses will be performed using SPSS 20.0 or higher.
9. Administrative aspects, monitoring and publication The investigator will preserve confidentiality of all subjects taking part in the study, in accordance with GCP and local regulations. The investigator must ensure that the subjects anonymity is maintained. Al data and material from one individual subject will be coded by an unique identification code. The key to the code is maintained by the investigator and research nurses. The validated data management system Castor will be used for data handling, according to GCP. Data will be stored for 15 years. Human material will be stored for 10 years. Source document and database verification will be performed by an independent monitor, according to a predefined monitoring plan. There will be minimal monitoring, once per year, as the study is judged to cause only marginal potential risk to the participants.
10. Public disclosure and publication policy This study has been made possible by an unrestricted grant from European Pharma Group (EPG), division Needle Free Insulin Products, the manufacturer of the InsujetTM jet-injector. EPG was not involved in the study design or writing of the protocol and will also not be involved in conducting the study, analysis of the data, presentation of the results, writing of the manuscript and the decision to submit for publication.

ELIGIBILITY:
Inclusion criteria

* Age 18-50 years
* Body-Mass Index 18-32 kg/m2
* Blood pressure <160/90 mmHg

Exclusion criteria

* Inability to provide informed consent
* Chronic use of medication other than oral contraceptives or thyroid hormone replacement therapy (with stable euthyroidism for at least 3 months)
* Treatment with systemic corticosteroids, immunosuppressive or cytostatic drugs
* Known allergy to aspart insulin
* History of a major cardiovascular disease event (myocardial infarction, stroke, symptomatic peripheral artery disease, coronary bypass surgery, percutaneous coronary or peripheral artery angioplasty) in the previous 6 months
* Presence of any other medical condition that might interfere with the study protocol
* Pregnancy or the intention to become pregnant
* Anemia, defined as an Hb of <8.1 mmol/l for male subjects and <7.5 for female subjects

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2015-02; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
(TmaxGIR) | 0-6 hrs
  The variability in time until maximal glucose lowering effect, as determined by exogenous glucose requirement (TmaxGIR) to maintain normoglycemia, after insulin injection. Primary endpoint of main study
Tmax (min) | 0-6 hrs
  Time to maximal exogenous glucose infusion rate (GIR, in ml/min/kg) required to maintain euglycaemia. Primary endpoint of sub study.

SECONDARY OUTCOMES:
CmaxGIR (mg/min) | 0-6 hrs
  Maximal GIR during the 6-hour study (from timepoint 0)
CmaxINS (pmol/l) | 0-6 hrs
  Maximal insulin concentration during the 6-hour study (from timepoint 0)
TmaxINS (min) | 0-6 hrs
  Time to maximal insulin concentration (Cmax)
AUCINS (pmol/min/l) | 0-6 hrs
  area under the insulin concentration curve during the 6-hour study
AUCGIR (g): | 0-6 hrs
  Area under the GIR curve during the 6-hour study (from timepoint 0)
T-GIRAUC50% (min) | 0-6 hrs
  Time of 50% of glucose disposal, i.e. the median of the GIR profile
T-INSAUC50% (min) | 0-6 hrs
  Time until 50% of insulin absorption (mean residence time, MRT)

OTHER OUTCOMES:
Tolerability | at second test day, at timepoint 0, for 5 minutes,
  The amount of discomfort or pain with the two administration methods using a numeric rating scale from 0 to 10 (VAS-score)

CONTACTS AND LOCATIONS:
Overall Officials: Bastiaan E de Galan, MD, PhD, Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboud university medical center, Nijmegen, Netherlands

REFERENCES:
- [Background] Mitragotri S. Current status and future prospects of needle-free liquid jet injectors. Nat Rev Drug Discov. 2006 Jul;5(7):543-8. doi: 10.1038/nrd2076. PMID 16816837
- [Background] Malone JI, Lowitt S, Grove NP, Shah SC. Comparison of insulin levels after injection by jet stream and disposable insulin syringe. Diabetes Care. 1986 Nov-Dec;9(6):637-40. doi: 10.2337/diacare.9.6.637. PMID 3542456
- [Background] Weller C, Linder M. Jet injection of insulin vs the syringe-and-needle method. JAMA. 1966 Mar 7;195(10):844-7. doi: 10.1001/jama.1966.03100100096027. PMID 12608170
- [Background] Taylor R, Home PD, Alberti KG. Plasma free insulin profiles after administration of insulin by jet and conventional syringe injection. Diabetes Care. 1981 May-Jun;4(3):377-9. doi: 10.2337/diacare.4.3.377. PMID 7047114
- [Background] Pehling GB, Gerich JE. Comparison of plasma insulin profiles after subcutaneous administration of insulin by jet spray and conventional needle injection in patients with insulin-dependent diabetes mellitus. Mayo Clin Proc. 1984 Nov;59(11):751-4. doi: 10.1016/s0025-6196(12)65585-2. PMID 6387316
- [Background] Halle JP, Lambert J, Lindmayer I, Menassa K, Coutu F, Moghrabi A, Legendre L, Legault C, Lalumiere G. Twice-daily mixed regular and NPH insulin injections with new jet injector versus conventional syringes: pharmacokinetics of insulin absorption. Diabetes Care. 1986 May-Jun;9(3):279-82. doi: 10.2337/diacare.9.3.279. PMID 3525057
- [Background] Kerum G, Profozic V, Granic M, Skrabalo Z. Blood glucose and free insulin levels after the administration of insulin by conventional syringe or jet injector in insulin treated type 2 diabetics. Horm Metab Res. 1987 Sep;19(9):422-5. doi: 10.1055/s-2007-1011842. PMID 3319860
- [Background] Lucas A, Ribas L, Salinas I, Audi L, Sanmarti A, Foz M. Insulin levels after injection by jet stream and disposable syringe. Diabetes Care. 1988 Mar;11(3):298-9. doi: 10.2337/diacare.11.3.298a. No abstract available. PMID 3046856
- [Background] Engwerda EE, Abbink EJ, Tack CJ, de Galan BE. Improved pharmacokinetic and pharmacodynamic profile of rapid-acting insulin using needle-free jet injection technology. Diabetes Care. 2011 Aug;34(8):1804-8. doi: 10.2337/dc11-0182. Epub 2011 Jun 29. PMID 21715522
- [Background] Gill GV, Yudkin JS, Keen H, Beran D. The insulin dilemma in resource-limited countries. A way forward? Diabetologia. 2011 Jan;54(1):19-24. doi: 10.1007/s00125-010-1897-3. Epub 2010 Sep 12. PMID 20835860
- [Background] Julious SA. Sample sizes for clinical trials with normal data. Stat Med. 2004 Jun 30;23(12):1921-86. doi: 10.1002/sim.1783. PMID 15195324
- [Derived] Engwerda EEC, Tack CJ, de Galan BE. Pharmacokinetic and Pharmacodynamic Variability of Insulin When Administered by Jet Injection. J Diabetes Sci Technol. 2017 Sep;11(5):947-952. doi: 10.1177/1932296817699638. Epub 2017 Mar 17. PMID 28303726